CLINICAL TRIAL: NCT06021327
Title: Comparison Of The Analgesic Effect Of Ultrasound-Guided Erector Spinae Plane Block And Ultrasound-Guided Retrolaminar Block In Patients Undergoing Video Assisted Thoracoscopic Surgery: A Prospective, Randomized Study.
Brief Title: Comparison Between Erector Spinae Plane Block And Retrolaminar Block In Patients Undergoing VATS.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam M Sayed, i.sharr866@gmail.com, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-327-2022
Record Dates: First submitted 2023-06-17; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Post-operative Analgesia; Retrolaminar Block; Erector Spinae Plan Block; VATS
Keywords: RLB; ESPB; VATS

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients will be randomized using a computer-generated list of random numbers, which will be sealed in closed envelopes. Patients will be randomly allocated to one of two groups; Group I (E) will receive a US-guided ESPB, while Group II (R) will receive a US-guided RLB. An anesthesiologist who is not involved in the data collection team will perform all nerve blocks. Intra- and postoperative data will be collected by an anesthesiologist or intensivist who is blinded to the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector spinae plane block (Active Comparator): will receive a US-guided ESPB
  Interventions: Procedure: Erector spinae plane block
- Retrolaminar block (Active Comparator): will receive a US-guided RLB
  Interventions: Procedure: Retrolaminar block

INTERVENTIONS:
Procedure: Erector spinae plane block — Under aseptic precautions, the ultrasound transducer will be placed on the patient's back in a longitudinal paramedian orientation approximately 3 cm from the midline. A short-bevel, 80 mm 22-gauge insulated nerve block needle will be inserted using an in-plane approach to contact the tip of the T4 transverse process , After negative aspiration of blood, a total of 20 mL of 0.25% bupivacaine will be injected through the needle. Adequacy of the block will be confirmed by ultrasonographic visualization of fluid spread (seen as a lifting of the erector spina muscles in both block) and after 15 min, documenting the sensory blockade will be done by using a piece of ice or cold object. If the desired sensory level fails to be achieved (T4 - T8), patients will be excluded from the study.
  Arms: Erector spinae plane block
Procedure: Retrolaminar block — Under aseptic precautions, the ultrasound transducer will be placed on the patient's back in a longitudinal paramedian orientation approximately 1 cm from the midline. A short-bevel, 80 mm 22-gauge insulated nerve block needle will be inserted using an in-plane approach to contact T4 lamina of the vertebra , After negative aspiration of blood, a total of 20 mL of 0.25% bupivacaine will be injected through the needle. And after 15 min, documenting the sensory blockade will be done by using a piece of ice or cold object. If the desired sensory level fails to be achieved (T4 - T8), patients will be excluded from the study.
  Arms: Retrolaminar block

SUMMARY:
Post-Video-assisted thoracoscopic surgery pain is a challenging clinical problem that may be associated with increased morbidity and mortality. The current study tests two techniques of regional anaesthesia to control post Video-assisted thoracoscopic surgery pain

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) is increasingly being used to manage primary lung cancer and helps reduce postoperative pain. However, it is a fact that pain following VATS can be severe and long-lasting. According to previous study, 18.8% of patients who undergo VATS present with persistent pain 2 months after surgery .The provision of pain relief is a significant consideration, and thoracic epidural analgesia is often regarded to be the gold standard. However, epidural analgesia is not always ideal, and other practical regional methods of analgesia after VATS have been proposed as Erector Spinae Plane Block (ESPB) or retrolaminar block (RLB) .

The retrolaminar block (RLB) is a modified paravertebral block that administers local anesthetic between the lamina of the thoracic vertebra and the erector spinal muscles, using landmark technique or under ultrasound guidance. Previous clinical study reported that RLB provides a good analgesic effect after VATS but was inferior to para-vertebral block(PVB).

Erector spinae plane block (ESPB) is a relatively new interfascial block procedure first described for thoracic analgesia. Previous clinical studies reported that ESPB provides a good analgesic effect after VATS (comparable with PVB) and decreases morphine consumption after Lateral thoracotomy surgery. Thus, anaesthesiologists now have a greater choice for regional anaesthesia for thoracic analgesia. Although ESPB and RLB have similar puncture sites, Only one clinical study comparing ESPB and RLB in breast surgery has been reported , The mentioned study was also limited only to female patients. both blocks were compared with PVB but There is no clinical study that compares ESPB and RLB directly in VATS. Although the mechanisms of action of both ESPB and RLB have not yet been completely clarified, one cadaveric study indicated that ESPB leads to a broader spread of the local analgesic into a more extensive range of intercostal spaces from a single point of injection than RLB . Another cadaveric study reported that the lateral pathway, which is involved in the blockade of the intercostal nerve or the lateral cutaneous branches of the intercostal nerves, is the primary mechanism of ESPB, in contrast to RLB.

Based on these anatomical studies, we hypothesize that ESPB can be superior to RLB for postoperative analgesia after VATS.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status class (ASA) I, II and III
* Patients undergoing VATS.

Exclusion Criteria:

1. Patient refusal
2. Coagulopathy, bleeding disorders,
3. In-ability to postpone anti-coagulation medications.
4. infection at the injection site
5. pregnancy, breastfeeding,
6. severe obesity (body mass index > 35 kg/m2 )
7. allergy to any drug used in the study
8. preoperative daily use of a non-steroidal anti-inflammatory drug (NSAID) or opioids,
9. Previous surgery in the thoracic vertebral region
10. Liver dysfunction.
11. Injury or a lesion at the block site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Total amount of morphine consumption in milligram in the first 24-hour postoperative in the two groups | 24-hour
  ESPB compared to RLB for postoperative analgesia after VATS

SECONDARY OUTCOMES:
• Time is required to perform the technique in minutes. | intraoperative
  between the start of US scanning and the local anesthetic injection
Heart Rate | intraoperative and 24 hours postoperative
  Heart rate (Bpm) at15 minutes after blocks are done before the induction (baseline), immediately after intubation, every 10 minutes intraoperative, immediately after extubation, and every 4 hour in the ICU for the first 24 hours.
Systolic arterial blood pressure | intraoperative and 24 hours postoperative
  Systolic arterial blood pressure in millimetre mercury at15 minutes after blocks are done before the induction (baseline), immediately after intubation, every 10 minutes intraoperative, immediately after extubation, and every 4 hour in the ICU for the first 24 hours.
Diastolic arterial blood pressure | intraoperative and 24 hours postoperative
  Diastolic arterial blood pressure in millimetre mercury at15 minutes after blocks are done before the induction (baseline), immediately after intubation, every 10 minutes intraoperative, immediately after extubation, and every 4 hour in the ICU for the first 24 hours.
Mean arterial blood pressure | intraoperative and 24 hours postoperative
  Mean arterial blood pressure in millimetre mercury at15 minutes after blocks are done before the induction (baseline), immediately after intubation, every 10 minutes intraoperative, immediately after extubation, and every 4 hour in the ICU for the first 24 hours.
• Intraoperative cardioactive drug use | Intraoperative
  The number of patients requiring ephedrine and atropine
• Intraoperative analgesics | Intraoperative
  The number of patients requiring additional doses of fentanyl. Total intraoperative IV fentanyl dose (above the standard two microgram / kilogram )
• Pain score according to VAS score | 24 hours
  VAS value obtained from the patient immediately after recovery from anesthesia then every 4 hours during the first 24 hours postoperatively.
• First request of analgesia postoperative | 24 hours Postoperative
  The elapsed time from the block procedure until the administration of the first postoperative rescue analgesia in hours
• Incidence of side effects related to opioid use | 24 hours Postoperative
  (postoperative nausea and vomiting (PONV), constipation, pruritus, urinary retention) in postoperative time.
• Incidence of complications or side-effects related to the block | 24 hours
  (bradycardia, hypotension, hematoma formation or intravascular injection).

CONTACTS AND LOCATIONS:
Overall Officials: Islam M Sayed, MS, Principal Investigator — Cairo University
Locations (1):
- Facalty of Medicine - Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Falcoz PE, Puyraveau M, Thomas PA, Decaluwe H, Hurtgen M, Petersen RH, Hansen H, Brunelli A; ESTS Database Committee and ESTS Minimally Invasive Interest Group. Video-assisted thoracoscopic surgery versus open lobectomy for primary non-small-cell lung cancer: a propensity-matched analysis of outcome from the European Society of Thoracic Surgeon database. Eur J Cardiothorac Surg. 2016 Feb;49(2):602-9. doi: 10.1093/ejcts/ezv154. Epub 2015 Apr 26. PMID 25913824
- [Background] Landreneau RJ, Mack MJ, Hazelrigg SR, Naunheim K, Dowling RD, Ritter P, Magee MJ, Nunchuck S, Keenan RJ, Ferson PF. Prevalence of chronic pain after pulmonary resection by thoracotomy or video-assisted thoracic surgery. J Thorac Cardiovasc Surg. 1994 Apr;107(4):1079-85; discussion 1085-6. doi: 10.1097/00132586-199412000-00051. PMID 8159030
- [Background] Homma T, Doki Y, Yamamoto Y, Ojima T, Shimada Y, Kitamura N, Yoshimura N. Risk factors of neuropathic pain after thoracic surgery. J Thorac Dis. 2018 May;10(5):2898-2907. doi: 10.21037/jtd.2018.05.25. PMID 29997955
- [Background] Crumley S, Schraag S. The role of local anaesthetic techniques in ERAS protocols for thoracic surgery. J Thorac Dis. 2018 Mar;10(3):1998-2004. doi: 10.21037/jtd.2018.02.48. PMID 29707356
- [Background] Shim JG, Ryu KH, Kim PO, Cho EA, Ahn JH, Yeon JE, Lee SH, Kang DY. Evaluation of ultrasound-guided erector spinae plane block for postoperative management of video-assisted thoracoscopic surgery: a prospective, randomized, controlled clinical trial. J Thorac Dis. 2020 Aug;12(8):4174-4182. doi: 10.21037/jtd-20-689. PMID 32944329
- [Background] Pfeiffer G, Oppitz N, Schone S, Richter-Heine I, Hohne M, Koltermann C. [Analgesia of the axilla using a paravertebral catheter in the lamina technique]. Anaesthesist. 2006 Apr;55(4):423-7. doi: 10.1007/s00101-005-0969-0. German. PMID 16404582
- [Background] Wang Q, Wei S, Li S, Yu J, Zhang G, Ni C, Sun L, Zheng H. Comparison of the analgesic effect of ultrasound-guided paravertebral block and ultrasound-guided retrolaminar block in Uniportal video-assisted Thoracoscopic surgery: a prospective, randomized study. BMC Cancer. 2021 Nov 16;21(1):1229. doi: 10.1186/s12885-021-08938-7. PMID 34784889
- [Background] Taketa Y, Irisawa Y, Fujitani T. Comparison of ultrasound-guided erector spinae plane block and thoracic paravertebral block for postoperative analgesia after video-assisted thoracic surgery: a randomized controlled non-inferiority clinical trial. Reg Anesth Pain Med. 2019 Nov 8:rapm-2019-100827. doi: 10.1136/rapm-2019-100827. Online ahead of print. PMID 31704789
- [Background] Chen N, Qiao Q, Chen R, Xu Q, Zhang Y, Tian Y. The effect of ultrasound-guided intercostal nerve block, single-injection erector spinae plane block and multiple-injection paravertebral block on postoperative analgesia in thoracoscopic surgery: A randomized, double-blinded, clinical trial. J Clin Anesth. 2020 Feb;59:106-111. doi: 10.1016/j.jclinane.2019.07.002. Epub 2019 Jul 19. PMID 31330457
- [Background] Macaire P, Ho N, Nguyen T, Nguyen B, Vu V, Quach C, Roques V, Capdevila X. Ultrasound-Guided Continuous Thoracic Erector Spinae Plane Block Within an Enhanced Recovery Program Is Associated with Decreased Opioid Consumption and Improved Patient Postoperative Rehabilitation After Open Cardiac Surgery-A Patient-Matched, Controlled Before-and-After Study. J Cardiothorac Vasc Anesth. 2019 Jun;33(6):1659-1667. doi: 10.1053/j.jvca.2018.11.021. Epub 2018 Nov 19. PMID 30665850
- [Background] Sotome S, Sawada A, Wada A, Shima H, Kutomi G, Yamakage M. Erector spinae plane block versus retrolaminar block for postoperative analgesia after breast surgery: a randomized controlled trial. J Anesth. 2021 Feb;35(1):27-34. doi: 10.1007/s00540-020-02855-y. Epub 2020 Sep 11. PMID 32915300
- [Background] Adhikary SD, Bernard S, Lopez H, Chin KJ. Erector Spinae Plane Block Versus Retrolaminar Block: A Magnetic Resonance Imaging and Anatomical Study. Reg Anesth Pain Med. 2018 Oct;43(7):756-762. doi: 10.1097/AAP.0000000000000798. PMID 29794943
- [Background] Ivanusic J, Konishi Y, Barrington MJ. A Cadaveric Study Investigating the Mechanism of Action of Erector Spinae Blockade. Reg Anesth Pain Med. 2018 Aug;43(6):567-571. doi: 10.1097/AAP.0000000000000789. PMID 29746445
- [Background] Onishi E, Toda N, Kameyama Y, Yamauchi M. Comparison of Clinical Efficacy and Anatomical Investigation between Retrolaminar Block and Erector Spinae Plane Block. Biomed Res Int. 2019 Mar 28;2019:2578396. doi: 10.1155/2019/2578396. eCollection 2019. PMID 31032339
- [Background] Pfizer Labs I, fda, cder. HIGHLIGHTS OF PRESCRIBING INFORMATION These highlights do not include all the information needed to use ROZLYTREK. 2019;(4):1-23. Available from: http://www.fda.gov/CompanionDiagnostics%0Ahttp://www.accessdata.fda.gov/drugsatfda_docs/label/2012/202570s002lbl.pdf
- [Background] Luo D, Wan X, Liu J, Tong T. Optimally estimating the sample mean from the sample size, median, mid-range, and/or mid-quartile range. Stat Methods Med Res. 2018 Jun;27(6):1785-1805. doi: 10.1177/0962280216669183. Epub 2016 Sep 27. PMID 27683581
- [Background] Wan X, Wang W, Liu J, Tong T. Estimating the sample mean and standard deviation from the sample size, median, range and/or interquartile range. BMC Med Res Methodol. 2014 Dec 19;14:135. doi: 10.1186/1471-2288-14-135. PMID 25524443

DOCUMENTS (1):
  • Study Protocol (2022-11-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT06021327/Prot_000.pdf